CLINICAL TRIAL: NCT05891119
Title: A Phase 1, Open-label, Drug-Drug Interaction Study to Investigate the Effect of Rocatinlimab (AMG 451) on the Pharmacokinetics of Multiple CYP450 Substrates in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Study to Investigate the Effect of Rocatinlimab (AMG 451) on the Pharmacokinetics of Multiple Cytochrome P450 (CYP450) Substrates in Participants With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20210147
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: Moderate to Severe Atopic Dermatitis; Rocatinlimab; AMG 451; Cytochrome P450 (CYP450) Substrates
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Caffeine; caffeine citrate; Metoprolol; Midazolam; Warfarin; Vitamin K; Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rocatinlimab and CYP450 Substrates (Experimental): A single oral dose of a CYP450 substrates cocktail which will include caffeine, metoprolol, midazolam, warfarin (with vitamin K), and omeprazole will be administered on Day 1.
  A single dose of rocatinlimab will then be administered on Days 8, 22, 36, 64, and 92.
  A single oral dose of CYP450 substrates cocktail in combination with a single dose of rocatinlimab will then be administered on Day 120.
  Interventions: Dietary Supplement: Caffeine; Drug: Metoprolol; Drug: Midazolam; Drug: Warfarin; Dietary Supplement: Vitamin K; Drug: Omeprazole; Drug: Rocatinlimab

INTERVENTIONS:
Dietary Supplement: Caffeine — Oral liquid
  Other Names: Caffeine Citrate
Drug: Metoprolol — Oral tablet
  Other Names: Metoprolol Tartrate
Drug: Midazolam — Oral liquid
  Other Names: Midazolam Hydrochloride
Drug: Warfarin — Oral tablet
  Other Names: Warfarin Sodium
Dietary Supplement: Vitamin K — Oral tablet
Drug: Omeprazole — Oral capsule
  Other Names: Omeprazole magnesium
Drug: Rocatinlimab — Subcutaneous injection
  Other Names: AMG 451

SUMMARY:
The primary objective of the study is to evaluate the pharmacokinetics (PK) of multiple cytochrome P450 (CYP450) substrates alone and in combination with rocatinlimab in participants with moderate to severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participant, aged 18 to 65 years
2. Diagnosis of AD, defined as diagnosis of AD for at least 6 months before signing of informed consent
3. Eczema Area Severity Index score ≥8 at the screening and Check-in
4. Investigator's Global Assessment (IGA) score ≥3 (on the 0 to 4 IGA scale) at screening and Check-in
5. ≥7% Body Surface Area of AD involvement at initial screening
6. History of inadequate response to topical corticosteroid therapy (TCS) of medium to higher potency within 6 months (with or without topical calcineurin inhibitors [TCI]) or for whom topical treatments are otherwise medically inadvisable (eg, because of important side effects or safety risks).
7. Provide signed informed consent

Exclusion Criteria:

1. Have previously completed or withdrawn from this study or any other study investigating rocatinlimab or have previously received a dose of an investigational drug within the past 90 days or 5 half-lives, whichever is longer, prior to Check-in
2. The use of any of the following treatments within 4 weeks before Check-in:

   * Systemic corticosteroids
   * Immunosuppressive/immunomodulating drugs
3. The use of any of the following treatments within one week before Check-in:

   1. Topical corticosteroids of any super-high potency
   2. Topical phosphodiesterase 4 (PDE4) inhibitors
   3. Phototherapy
4. Administration, within 14 days before baseline or within a period of 5 times the elimination half-life of the medication before baseline, whichever is longer, of any medication that is a known inducer or inhibitor of either one or more of the following cytochrome P450 (CYP) enzymes: CYP3A4, CYP2C19, CYP2C9, CYP2D6, and CYP1A2. Participants who are on any of these medications at the time of screening and cannot be safely taken off these medications will be excluded from the study.
5. Any contraindication to one or more of the following drugs, according to the applicable labeling:

   * Midazolam
   * Omeprazole
   * Warfarin (and Vitamin K)
   * Caffeine
   * Metoprolol
6. Consumption of any 1 or more of the following food items and/or beverages within 1 week prior to Check-in:

   * Grapefruit or grapefruit juice, apple or apple juice, orange or orange juice, lemons or lemon juice, limes or lime juice
   * Vegetables from the mustard green family (eg, broccoli)
   * Charbroiled meats
   * Caffeinated beverages, foods or drugs containing caffeine
7. History of alcoholism or drug/chemical abuse within 1 year prior to Check-in or regular alcohol consumption (>14 units per week for males and >7 units for females)
8. Smoke more than 10 cigarettes or use the equivalent (as determined by site staff) tobacco- or nicotine-containing products per day and unwilling to adhere to smoking restrictions.
9. Poor metabolizers for CYP2C9, CYP2C19, or CYP2D6 based on genotyping
10. Presence of any one or more of the following lab abnormalities at screening or Check-in:

    • Platelet count <100k /µL, international normalized ratio (INR)>1.2, prothrombin time (PT)>13.5 sec or partial thromboplastin time (PTT)>35 sec
11. Active, chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiprotozoals, or antifungals at screening or Check-in
12. Superficial skin infections, including tinea infections, within 2 weeks prior to Check-in
13. History of acquired, common variable, primary or secondary immunodeficiency
14. Positive hepatitis B or hepatitis C panel and/or positive human immunodeficiency virus test, at screening as per Center for Disease Control interpretation. Participants whose hepatitis B and C results are compatible with prior immunity (resulting from inoculation) may be included. Participants with positive hepatitis B core antibody will be excluded.
15. Active malignancy, multiple myeloma, myeloproliferative or lymphoproliferative disorder, or a history of any of these conditions within 5 years prior to informed consent (except curatively treated in situ cervical carcinoma, cutaneous basal cell carcinoma, or cutaneous squamous cell carcinoma)
16. Diagnosis of a helminth parasitic infection within 6 months prior to screening that had not been treated with or failed to respond to standard of care therapy.
17. History of suicidal ideation (thoughts), suicide-related behaviors, suicide attempt(s), depression or major psychiatric illness within 6 months prior to signing the informed consent
18. Female participants who are pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study through 18 weeks after the end of study visit
19. Unwilling to adhere to contraceptive requirements through 18 weeks after the end of study visit
20. Male participant with a pregnant partner or partner planning to become pregnant while the participant is on study through 18 weeks after the end of study visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-06-03 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of CYP450 Substrate | Day 1
Cmax of CYP450 Substrate | Day 120
Area Under the Serum Concentration-Time Curve from Time Zero to Time of Last Quantifiable Concentration (AUClast) of CYP450 Substrate | Day 1
AUClast of CYP450 Substrate | Day 120
Area Under the Serum Concentration-Time Curve from Time Zero to Infinity (AUCinf) of CYP450 Substrate | Day 1
AUCinf of CYP450 Substrate | Day 120

SECONDARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to Day 238
Number of Participants with Serious Adverse Events (SAEs) | Up to Day 238
Number of Participants with Anti-rocatinlimab Antibody Formation | Up to Day 238

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- United States (7):
  - Velocity Clinical Research, North Hollywood, North Hollywood, California
  - Accel Research Sites (ACR), DeLand, Florida
  - Direct Helpers Research Center (DHRC), Hialeah, Florida
  - Axis Clinicals, LCC, Dilworth, Minnesota
  - DermDox Dermatology Centers, PC - Camp Hill, Camp Hill, Pennsylvania
  - Velocity Clinical Research -Spartanburg, Spartanburg, South Carolina
  - DermDox Dermatology Centers, PC - Sugarloaf, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com